CLINICAL TRIAL: NCT05714761
Title: Postpartum Dysglycemia Screening With Continuous Glucose Monitoring
Brief Title: Postpartum Continuous Glucose Monitoring (CGM) Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: DexCom, Inc. (Industry)
Responsible Party: Principal Investigator, Grenye O'Malley, Assistant Professor, Icahn School of Medicine at Mount Sinai
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: STUDY-20-02062
Record Dates: First submitted 2023-01-27; First posted 2023-02-06 (Actual); Results first posted 2025-03-20 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Gestational Diabetes
Keywords: gestational diabetes; oral glucose tolerance test; glucose sensor
MeSH Terms: conditions — Diabetes, Gestational

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Postpartum glucose sensor (Other): Will wear glucose sensor for 10 days postpartum and at time of glucose tolerance test.
  Interventions: Device: Dexcom glucose sensor

INTERVENTIONS:
Device: Dexcom glucose sensor — Use of a Dexcom G6 Pro

SUMMARY:
This research study is being done to assess if using a glucose sensor (also known as a continuous glucose monitor) after childbirth can help identify women who are at risk of developing diabetes after having diabetes during pregnancy or gestational diabetes. Currently, screening for diabetes after childbirth is performed with an oral glucose tolerance test 6-12 weeks after delivery, but this is burdensome. This study will use a glucose sensor worn on the skin for 10 days. The data from the sensor will be compared to the standard oral glucose tolerance test. This is a single site study at the Icahn School of Medicine at Mount Sinai. The research team plans to enroll 50 participants aged 18years or older into the study. Participation in the study is expected to last up to 20 weeks and involves 4-5 visits depending on if enrollment is in the 3rd trimester of pregnancy or immediate postpartum. Study procedures include 1. Consent & screening. 2.Sensor placement and download after 10 days of wear. 3. a second sensor placement 2-5 days before oral glucose tolerance test (OGTT).

ELIGIBILITY:
Inclusion criteria:

* include diagnosis of gestational diabetes during a current or recent pregnancy
* age 18 or older.

Exclusion criteria:

* include known pregestational diabetes,
* known skin adhesive allergy which would prevent subject from wearing a CGM,
* chronic glucocorticoid use which is planned to be ongoing after labor and delivery discharge.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2023-02-16 (Actual); Primary Completion 2024-03-08 (Actual); Study Completion 2024-03-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Grenye O'Malley, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (1):
- Icahn School of Medicine at Mount Sinai, New York, New York, United States

IPD SHARING:
Plan to Share IPD: No
Aggregate data will be reported

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment was conducted from February 2023-January 2024 at a single urban medical center.
Groups:
- Postpartum Glucose Sensor: Glucose sensor worn for up to 10 days postpartum and at time of glucose tolerance test.
  Dexcom glucose sensor: Use of a Dexcom G6 Pro
Period: Overall Study
Arm/Group | Postpartum Glucose Sensor
Started | 50
CGM Returned | 43
Completed Routine Postpartum Oral Glucose Tolerance Test (OGTT) | 34
Returned the Second CGM Sensor | 30
Completed | 30
Not Completed | 20
Not completed — Lost to Follow-up | 3
Not completed — Withdrawal by Subject | 3
Not completed — unblinding of sensor data | 1
Not completed — did not complete routine postpartum OGTT | 9
Not completed — did not return second CGM sensor | 4

BASELINE CHARACTERISTICS:
Arm/Group | Postpartum Glucose Sensor
Number analyzed (Participants) | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 36 (5.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50
  Male | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 20
  Non-Hispanic Black | 12
  Asian | 11
  Hispanic | 7
Pre-pregnancy body mass index [Median (Inter-Quartile Range); unit: kg/m^2] | 26.6 [23.8 to 30.5]
Insurance type [Count of Participants; unit: Participants]
  Commercial | 33
  Medicaid | 17
Education Level [Count of Participants; unit: Participants]
  Some high school or less | 7
  High school/GED | 3
  Some college | 8
  College degree | 16
  Post college | 14
  Prefer not to answer | 2
Family history of type 2 diabetes [Count of Participants; unit: Participants] | 30
Multigravida [Count of Participants; unit: Participants] | 39
Gestational diabetes (GDM) in prior pregnancy [Count of Participants; unit: Participants] | 13
Number of prenatal visits [Mean (Standard Deviation); unit: visits] | 13.8 (4.6)
GDM management [Count of Participants; unit: Participants]
  Diet/Lifestyle only | 23
  Oral agents | 4
  Insulin | 23
Hypertensive complications [Count of Participants; unit: Participants] | 11
Delivery type [Count of Participants; unit: Participants]
  Vaginal | 33
  C-section | 17

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With at Least 72 Hours of CGM Data Downloaded.
Description: Number of participants who returned first sensors and had at least 72 hours of CGM data downloaded.
Time Frame: Postpartum days 10-20
Measure: Count of Participants; unit: Participants
Arm/Group | Postpartum Glucose Sensor
Number analyzed (Participants) | 50
Participants | 43

2. Secondary Outcome: Specificity
Description: Specificity for CGM compared to oral glucose tolerance test for diagnosis of diabetes, impaired glucose tolerance and impaired fasting glucose. The specificity of a test is the number and proportion of people who test negative among all those who actually do not have that disease. A higher specificity in a test indicates it is better at correctly identifying individuals with the condition.
  Specificity for Time in Range 70-180 mg/dL of <96% for abnormal OGTT is reported.
Time Frame: up to 12 weeks postpartum
Population: Results for usable data
Measure: Number; unit: percent
Groups:
- Postpartum Glucose Sensor: Glucose sensor worn postpartum days 1-13 and at time of glucose tolerance test.
  Dexcom glucose sensor: Use of a Dexcom G6 Pro
- Second Sensor: Participants given a second sensor at 6 weeks after pregnancy complicated by GDM and worn at home for up to 10 days at time of glucose tolerance test. Data collected for 4-12 weeks postpartum.
Arm/Group | Postpartum Glucose Sensor | Second Sensor
Number analyzed (Participants) | 34 | 29
percent | 78 | 83.33

3. Secondary Outcome: Sensitivity
Description: Sensitivity for CGM compared to oral glucose tolerance test for diagnosis of diabetes, impaired glucose tolerance and impaired fasting glucose. The sensitivity of a test is the number of people who test positive among all those who actually have the disease. A higher sensitivity in a test indicates it is better at correctly identifying those who have the condition and not missing cases.
  Sensitivity for Time in Range 70-180 mg/dL of <96% for abnormal OGTT is reported.
Time Frame: up to 12 weeks postpartum
Population: Results for usable data
Measure: Number; unit: percent
Groups:
- Second Sensor: Participants given a second sensor at 6 weeks after pregnancy complicated by GDM and worn at home for up to 10 days.
Arm/Group | Postpartum Glucose Sensor | Second Sensor
Number analyzed (Participants) | 34 | 29
percent | 100 | 66.67

4. Secondary Outcome: Positive Predictive Value (PPV)
Description: PPV for CGM compared to oral glucose tolerance test for diagnosis of diabetes, impaired glucose tolerance and impaired fasting glucose. Positive predictive value is the probability that following a positive test result, that individual will truly have that specific disease.
  Positive predictive value (PPV) of Time in Range 70-180 mg/dL of <96% to predict abnormal OGTT is reported.
Time Frame: up to 12 weeks postpartum
Measure: Number; unit: percent
Arm/Group | Postpartum Glucose Sensor | Second Sensor
Number analyzed (Participants) | 43 | 30
percent | 53.49 | 50

5. Secondary Outcome: Positive Likelihood Ratio (PLR)
Description: PLR for CGM compared to oral glucose tolerance test for diagnosis of diabetes, impaired glucose tolerance and impaired fasting glucose. PLR compares the likelihood of a positive test result in people with a disease to the likelihood in people without the disease and is used to help determine how likely a disease is present if a test is positive. The higher the PRL, the stronger the evidence that a positive test result supports the presence of the condition.
  PLR of Time in Range 70-180 mg/dL of <96% to predict abnormal OGTT is reported.
Time Frame: up to 12 weeks postpartum
Measure: Number; unit: ratio
Arm/Group | Postpartum Glucose Sensor | Second Sensor
Number analyzed (Participants) | 43 | 30
ratio | 4.5 | 3.83

6. Secondary Outcome: Negative Predictive Value (NPV)
Description: NPV for CGM compared to oral glucose tolerance test for diagnosis of diabetes, impaired glucose tolerance and impaired fasting glucose. Negative predictive value is the probability that following a negative test result, that individual will truly not have that specific disease.
  NPV of Time in Range 70-180 mg/dL of <96% to predict abnormal OGTT is reported.
Time Frame: up to 12 weeks postpartum
Measure: Number; unit: percent
Arm/Group | Postpartum Glucose Sensor | Second Sensor
Number analyzed (Participants) | 43 | 30
percent | 100 | 90

7. Secondary Outcome: Negative Likelihood Ratio (NLR)
Description: NLR estimates how likely a patient is to not have a disease after a negative test. The lower the NRL, the stronger the evidence that a negative test result supports the absence of the condition.
  NLR of Time in Range 70-180 mg/dL of <96% to predict abnormal OGTT is reported.
Time Frame: up to 12 weeks postpartum
Measure: Number; unit: ratio
Arm/Group | Postpartum Glucose Sensor | Second Sensor
Number analyzed (Participants) | 43 | 30
ratio | 0 | 0.4

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | Postpartum Glucose Sensor | Second Sensor
All-Cause Mortality (participants affected / at risk) | 0/43 | 0/30
Serious Adverse Events (participants affected / at risk) | 0/43 | 0/30
Other Adverse Events (participants affected / at risk) | 0/43 | 0/30

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-12-21): https://cdn.clinicaltrials.gov/large-docs/61/NCT05714761/Prot_SAP_000.pdf